CLINICAL TRIAL: NCT06077227
Title: Immersive Healing: The Therapeutic Potential of Virtual Reality in Phantom Limb Experience
Brief Title: Immersive Healing: The Therapeutic Potential of Virtual Reality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00100006
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-08

CONDITIONS: Phantom Limb Pain (PLP)
Keywords: amputee; pain management; virtual reality (VR) therapy
MeSH Terms: conditions — Phantom Limb; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Pre- and post-intervention surveys will be used to assess the effects of virtual reality (VR) therapy on the phantom limb experience in the intervention group. Matched controls from the registry will be surveyed on their phantom limb symptoms at matching time intervals to the intervention group for comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Virtual Reality (VR) Intervention (Experimental): Individuals undergoing virtual reality therapy intervention
  Interventions: Device: virtual reality therapy
- Matched Control (Sham Comparator): The matched controls will receive standard care without the VR intervention
  Interventions: Other: matched control group

INTERVENTIONS:
Device: virtual reality therapy — 6 2 times weekly sessions of 30-minute VR therapy in the office with pre- and post-intervention surveys
  Other Names: VR Intervention
  Arms: Virtual Reality (VR) Intervention
Other: matched control group — taking the same surveys as the VR intervention group on a weekly basis for 6 weeks
  Other Names: control group
  Arms: Matched Control

SUMMARY:
Phantom limb pain (PLP) is a significant and pervasive issue among upper limb amputees, severely impacting their quality of life. The literature delineating prevalence of upper versus lower limb amputations is limited, but the prevalence of total amputations in the United States is estimated to reach 3 million individuals by 2050, with approximately 185,000 new cases annually. PLP affects 60-68% of these patients, leading to heightened levels of anxiety, depression, and reduced overall well-being.

DETAILED DESCRIPTION:
Although studies exploring the efficacy of VR therapy for PLP have reported positive outcomes, several limitations, such as small sample sizes, lack of randomization, and inconsistent treatment protocols, have impeded widespread adoption of these innovative approaches. Additionally, the literature does not sufficiently delineate which aspects of the phantom limb experience may be addressed with VR therapy. To overcome these limitations and optimize treatment efficacy, it is crucial to gain a comprehensive understanding of the phantom limb experience, including both somatosensory and kinesthesia-related symptoms. Additionally, this study will address these limitations by employing a larger sample size, rigorous methodology, and a standardized treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* History of major limb amputation
* Age > 18 years old
* Presence of phantom limb pain or negative phantom sensation(s)

Exclusion Criteria:

* Active mental illness, neurological disease, or cognitive impairment that would interfere with survey completion
* Those without phantom limb pain or negative phantom limb sensations
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Phantom limb pain levels using Short-form McGill Pain Questionnaire (SF-MPQ) | Baseline
  Short-form McGill Pain Questionnaire - The maximum score an individual can reach on the MPQ is 78. According to the questionnaire, a person with a score of 0 effectively does not experience pain. A person with a high score, nearer to the highest score of 78, more than likely deals with chronic pain daily.
Phantom limb pain levels using Short-form McGill Pain Questionnaire (SF-MPQ) | Week 1
  Short-form McGill Pain Questionnaire - The maximum score an individual can reach on the MPQ is 78. According to the questionnaire, a person with a score of 0 effectively does not experience pain. A person with a high score, nearer to the highest score of 78, more than likely deals with chronic pain daily.
Phantom limb pain levels using Short-form McGill Pain Questionnaire (SF-MPQ) | Week 2
  Short-form McGill Pain Questionnaire - The maximum score an individual can reach on the MPQ is 78. According to the questionnaire, a person with a score of 0 effectively does not experience pain. A person with a high score, nearer to the highest score of 78, more than likely deals with chronic pain daily.
Phantom limb pain levels using Short-form McGill Pain Questionnaire (SF-MPQ) | Week 3
  Short-form McGill Pain Questionnaire - The maximum score an individual can reach on the MPQ is 78. According to the questionnaire, a person with a score of 0 effectively does not experience pain. A person with a high score, nearer to the highest score of 78, more than likely deals with chronic pain daily.
Phantom limb pain levels using Short-form McGill Pain Questionnaire (SF-MPQ) | Week 6
  Short-form McGill Pain Questionnaire - The maximum score an individual can reach on the MPQ is 78. According to the questionnaire, a person with a score of 0 effectively does not experience pain. A person with a high score, nearer to the highest score of 78, more than likely deals with chronic pain daily.

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI) scores | Hour 24
  Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain - Scores range from 0 to 10 with higher scores indicating greater pain interference.
Change in Short-Form McGill Pain Questionnaire (SF-MPQ) scores | Week 6
  A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
  Consists of 22 different descriptors of pain and each item is rated based on a 0-10 scale with 0 equal to no pain and 10 equal to the worst pain ever during the past week. The total score is calculated by summing 22 individual scores.
Phantom Limb Experience Survey score | Baseline
  it is qualitative and there is no good or bad, this is just to define the population and better characterize phantom limb experience - assesses presence, onset, location, character, intensity, triggers, and treatment of phantom limb sensations and phantom limb pain. Includes questions on phantom limb posture, movement, size changes, and telescoping.
Change in Virtual Reality (VR) Therapy Survey scores | Week 6
  There are several questions within this survey to assess attitude towards VR, which activities are favored and then the effect VR had on them. There is a mix of qualitative questions and quantitative. Quantitative questions are on Likert Scale 1-5. An interval change of +1 on Likert scale would be "good" for question on posture, control over limb. For how long the therapy effect lasts after session is over, it will vary from hours to days to weeks (which is why all descriptors are in there). Even if it lasted 1 hour this would be considered "good".
System Usability Scale | Week 6
  Assesses subjective usability and satisfaction with the VR system - A perfect score of 100% signifies flawless usability and an exceptional user experience. The average SUS score is 68, and scores up to 70% are generally considered good; a good sus score indicates a decent level of usability.
Simulator Sickness Questionnaire | Week 6
  negligible (< 5), minimal (5 - 10), significant (10 - 15), and concerning (15 - 20) symptoms. A simulator resulting in total scores above 20 is considered "bad"
Change in EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) scores | Week 6
  Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Gaston, MD, Principal Investigator — Atrium Health Musculoskeletal Institute
Locations (1):
- OrthoCarolina Hand Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data that underlie the results reported in this article, after deidentification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal